CLINICAL TRIAL: NCT05620186
Title: Registry Endovascular Training Curriculum PROSPECT for Surgical Trainees (PROficiency-based StePwise Endovascular Curricular Training Program)
Brief Title: PROficiency Based StePwise Endovascular Curricular Training: Multicentric Registry
Acronym: PROSPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BC-877
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Vascular Diseases
Keywords: simulation based education; endovascular procedures
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Registry, no comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Original PROSPECT (Other): Original, distributed PROSPECT where trainees learn at their own pace in between, before/after clinical activities
  Interventions: Other: PROSPECT
- Massed PROSPECT (Other): Massed, bootcamp-style training form of PROSPECT where trainees are exempt from clinical duties
  Interventions: Other: PROSPECT

INTERVENTIONS:
Other: PROSPECT — PROficiency Based StePwise Endovascular Curricular Training

SUMMARY:
The goal of this multicentric registry is to gather data from trainees completing PROSPECT: a PROficiency Based StePwise Endovascular Curricular Training to obtain basic cognitive and technical skills. The main goals are to identify if:

* Results from a previous randomised controlled trail can be reproduced in real life.
* Evaluate skills retention after program completion.
* Assess real life implementation of the training program.

DETAILED DESCRIPTION:
A validated PROSPECT (PROficiency-based StePwise Endovascular Curricular Training) training has been integrated into the training of surgical residents to teach basic cognitive, technical and non-technical endovascular skills. The program uses virtual reality simulation and E-learning. During the four modules of the program, formative feedback is given after each training session. Only after achieving a predetermined benchmark score, trainees can progress to the next module.

Surgical trainees completing PROSPECT showed superior real live endovascular performance compared to the traditionally trained in a single centre randomised controlled trial (RCT). The curriculum was integrated locally, but also introduced in other centers: national and international. Local tutors teach the curriculum to trainees after standardized training on the modalities of PROSPECT by the researchers of the Ghent.

A registry is maintained and coordinated by the Ghent research group in which all educational data regarding this training is collected and processed anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Surgical trainee
* Knowledge and technical skill level evaluated
* Demographics questionnaire and general MCQ test completed
* Endovascular simulated exercise completed after familiarization with the simulator

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive skills | comparison before program start and after completion. This means through study completion.
  Multiple Choice Question test (min: 0, max: 20, the higher the score, the better)
Technical skills | comparison before program start and after completion. This means through study completion.
  Rating scale assessment and simulator metrics

SECONDARY OUTCOMES:
Cognitive skills retention | 3, 6 and 12 months after program completion
  Multiple Choice Question test (min: 0, max: 20, the higher the score, the better)
Technical skills retention | 3, 6 and 12 months after program completion
  Rating scale assessment and simulator metrics

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Van Herzeele, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - KU Leuven, Leuven
- CAMES, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No